CLINICAL TRIAL: NCT05363995
Title: Feasibility and Preliminary Effectiveness of a Blended E-health Intervention for Improving Sleep and the Biological Clock Among University Students (i-Sleep & BioClock)
Brief Title: Feasibility Trial i-Sleep & BioClock Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University (Other)
Responsible Party: Principal Investigator, Philip Spinhoven, Prof. Philip Spinhoven, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BioClockWP1.4
Record Dates: First submitted 2022-04-26; First posted 2022-05-06 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Insomnia
Keywords: sleep; biological clock; CBTi; e-health intervention; university students
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Single arm open feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Blended e-health intervention
  Interventions: Behavioral: i-Sleep & BioClock Intervention

INTERVENTIONS:
Behavioral: i-Sleep & BioClock Intervention — The 'i-Sleep & BioClock' intervention aims at improving sleep and the biological clock among university students. It is incorporates evidence-based techniques such as cognitive behavioural therapy for insomnia (CBTi). The intervention has a duration of 5 weeks and consists of five modules:
  1. psychoeducation on insomnia, sleep hygiene and the biological clock,
  2. stimulus control and sleep restriction therapy,
  3. worrying and relaxation exercises,
  4. cognitive therapy to change dysfunctional thoughts about sleep, and
  5. summary module, relapse prevention, and plan for the future.
  The intervention is supported by e-coaches who give personalized written feedback. Students will fill in a sleep & light exposure diary daily.

SUMMARY:
Students often suffer from sleep problems and circadian rhythm disruptions which affect their mental health and daily functioning. The aim of this project is to develop, implement and evaluate an e-health intervention that targets the biological clock and improves the sleep patterns of university students in order to prevent the development or exacerbation of mental health problems. The investigators will assess the feasibility, usability and acceptability of the intervention in this pilot trial.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the e-health modules, in terms of overall acceptability, feasibility, and usability. The secondary objective is to evaluate preliminary effectiveness on the outcomes mentioned below.

ELIGIBILITY:
Inclusion Criteria:

* Being fluent in Dutch and/or English
* Being enrolled as a student (Bachelor, Master or PhD) in one of the seven participating universities (Leiden University, Vrije Universiteit Amsterdam, Utrecht University, Maastricht University, Erasmus University Rotterdam, University of Amsterdam, Inholland University of Applied Sciences)
* Being ≥ 16 years old
* Having self-reported sleep problems; Insomnia Severity Index ≥ 8 (at least subthreshold insomnia)

Exclusion Criteria:

* Current risk for suicidal behaviour

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | Change from baseline (T0) to 7 weeks after baseline (T1)
  7-item self-report instrument to assess insomnia severity, scores 0-28, higher scores indicating more insomnia severity

SECONDARY OUTCOMES:
Sleep and light exposure diary | Change from week 0 (7 days prior to intervention period) to week 8 (7 days after T1)
  This diary includes measures such as sleep efficiency, sleep onset latency, total sleep time, wake after sleep onset, number of awakenings, early morning awakening, time spent outside, screen use before bedtime)
Munich Chronotype Questionnaire (MCTQ) | Change from baseline (T0) to 7 weeks after baseline (T1)
  Self-rated scale to assess individual phase of entrainment on work and work-free days, Addresses questions about: bedtime, time spent in bed awake before deciding to turn off the lights, how long it takes to fall asleep, wake up time, get up time on work and work-free days. MCTQ uses the midpoint between sleep on- and offset on free days (mid-sleep on free days, MSF) to assess chronotype
Patient Health Questionnaire (PHQ-9) | Change from baseline (T0) to 7 weeks after baseline (T1)
  9-items self-report instrument for severity of depressive symptoms, scores ranging from 0-27, higher scores indicating more severe depression
Generalised Anxiety Disorder scale (GAD-7) | Change from baseline (T0) to 7 weeks after baseline (T1)
  7-items self-report instrument for severity of anxiety symptoms, scores ranging from 0-21, higher scores indicating more severe anxiety
Work and Social Adjustment Scale (WSAS) | Change from baseline (T0) to 7 weeks after baseline (T1)
  5-item self-report instrument for impairment of functioning, scores ranging from 0-40, higher scores indicating more impairment in functioning
Mental Health Quality of Life questionnaire (MHQoL) | Change from baseline (T0) to 7 weeks after baseline (T1)
  7-item self report instrument for quality of life measure for use in people with mental health problems, scores ranging from 0-21, higher scores indicating higher quality of life, and MHQoL-VAS visual scale ranging from 0 (worst imaginable psychological wellbeing) to 10 (best imaginable psychological wellbeing)

OTHER OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | 7 weeks after baseline (T1)
  8-item self-report questionnaire for client satisfaction with services, total score ranging from 8-32, higher indicating higher satisfaction
System Usability Scale (SUS-10) | 7 weeks after baseline (T1)
  10-item self-report scale for system usability, five response options for respondents; from strongly agree to strongly disagree, scores ranging from 0-40, higher scores indicating better system usability
Working Alliance Inventory for guided Internet interventions (WAI-I) | 7 weeks after baseline (T1)
  12-item self-report instrument to capture alliance in guided Internet interventions, 5-point Likert scale ranging from 1 (never) to 5 (always), scores ranging from 12-60, higher scores indicating better alliance
Acceptability and usability of the sleep & light exposure diary | 7 weeks after baseline (T1)
  11 items on the sleep & light exposure diary, 5 point Likert Scale, scores ranging from 0-44, higher scores indicating better usability and acceptability, one visual scale on usefulness of the diary, 0 (not at all useful) to 10 (Very much useful)
Adherence to the program | Through study completion, on average 7 weeks
  Will be measured by the total number of completed modules and lessons, time spent in the platform, and the number of logins

CONTACTS AND LOCATIONS:
Overall Officials: Niki Antypa, PhD, Principal Investigator — Leiden University
Locations (1):
- Leiden Univeristy, Leiden, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pape LM, Antypa N, Spinhoven P, van Straten A, Struijs SY; Caring Universities Consortium. Open pilot study of a guided digital self-help intervention targeting sleep and the biological clock in university students using a pre-test post-test design. Sci Rep. 2025 Jul 1;15(1):21837. doi: 10.1038/s41598-025-04891-8. PMID 40593043